CLINICAL TRIAL: NCT02222948
Title: A Phase 2a/2b Double-Blind, Randomized, Placebo-Controlled Study Assessing Efficacy, Safety, and Dose-Response of Vatelizumab in Patients With Relapsing-Remitting Multiple Sclerosis (RRMS)
Brief Title: Efficacy and Safety of Vatelizumab in Patients With Relapsing-Remitting Multiple Sclerosis
Acronym: EMPIRE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued based on planned interim analysis of the primary endpoint. Not linked to any safety concern.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI13839; 2014-001643-20 (EudraCT Number); U1111-1153-3840 (Other: UTN)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vatelizumab Dose 1 (Experimental): Vatelizumab dose 1 at Weeks 0, 2, 4 and 8
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 2 (Experimental): Vatelizumab dose 2 at Weeks 0, 2, 4 and 8
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 3 (Experimental): Vatelizumab dose 3 at Weeks 0, 2, 4 and 8
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 4 (Experimental): Vatelizumab dose 4 at Weeks 0, 2, 4 and 8
  Interventions: Drug: Vatelizumab
- Placebo (Placebo Comparator): Placebo (for Vatelizumab) at Weeks 0, 2, 4 and 8
  Interventions: Drug: Placebo (for Vatelizumab)

INTERVENTIONS:
Drug: Vatelizumab — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: SAR339658
  Arms: Vatelizumab Dose 1; Vatelizumab Dose 2; Vatelizumab Dose 3; Vatelizumab Dose 4
Drug: Placebo (for Vatelizumab) — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Arms: Placebo

SUMMARY:
Primary Objectives:

* To assess the efficacy of vatelizumab compared to placebo as measured by a reduction in new contrast-enhancing lesions (CELs) in relapsing remitting multiple sclerosis (RRMS) patients.
* To evaluate multiple doses of vatelizumab for a dose-response.

Secondary Objectives:

* To evaluate the safety and tolerability of vatelizumab compared to placebo.
* To evaluate the pharmacokinetics (PK) of vatelizumab.

DETAILED DESCRIPTION:
The duration of study per patient will be up to 108 weeks, including a screening period of up to 4 weeks, a treatment period of 12 weeks and a post-treatment safety follow-up period of up to 92 weeks.

Patients completing the 12-week treatment period may enter an optional long-term extension study in which all subjects will receive vatelizumab.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of relapsing-remitting multiple sclerosis (RRMS). At least 1 documented relapse in the past 12 months. At least 1 contrast-enhancing lesion (CEL) on magnetic resonance imaging (MRI) in the past 12 months and/or at screening.

At least 3 T2 lesions on screening MRI.

Exclusion criteria:

Diagnosis of primary progressive or secondary progressive MS. Expanded disability status scale (EDSS) score >5.5. Relapse within 30 days prior to enrollment. Prior immunosuppressive treatment within protocol-specified time periods. Prior treatment with natalizumab (Tysabri®). History of bleeding/platelet disorders, malignancy, certain infections as defined in the protocol, or any other past or current medical conditions that would adversely affect the patient's participation in the study.

Pregnancy or breast-feeding. Other protocol-defined inclusion/exclusion criteria may apply.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reduction in the cumulative number of new contrast-enhancing lesions on MRI | from Week 4 to Week 12

SECONDARY OUTCOMES:
Safety: proportion of patients experiencing adverse events | up to Week 104
Pharmacokinetics: serum concentrations of vatelizumab | up to Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- United States (12):
  - Investigational Site Number 840004, Cullman, Alabama
  - Investigational Site Number 840009, Phoenix, Arizona
  - Investigational Site Number 840005, Fort Collins, Colorado
  - Investigational Site Number 840014, Washington D.C., District of Columbia
  - Investigational Site Number 840007, Ormond Beach, Florida
  - Investigational Site Number 840012, Tampa, Florida
  - Investigational Site Number 840001, Latham, New York
  - Investigational Site Number 840015, Knoxville, Tennessee
  - Investigational Site Number 840003, Round Rock, Texas
  - Investigational Site Number 840016, San Antonio, Texas
  - Investigational Site Number 840002, Salt Lake City, Utah
  - Investigational Site Number 840008, Seattle, Washington
- Canada (2):
  - Investigational Site Number 124001, Greenfield Park
  - Investigational Site Number 124002, Québec
- Poland (7):
  - Investigational Site Number 616008, Bydgoszcz
  - Investigational Site Number 616007, Lodz
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616004, Lublin
  - Investigational Site Number 616003, Lublin
  - Investigational Site Number 616002, Szczecin
  - Investigational Site Number 616006, Warsaw
- Russia (9):
  - Investigational Site Number 643010, Kazan'
  - Investigational Site Number 643009, Moscow
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643006, Nizhny Novgorod
  - Investigational Site Number 643005, Nizhny Novgorod
  - Investigational Site Number 643008, Novosibirsk
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg
- Sweden (2):
  - Investigational Site Number 752002, Gothenburg
  - Investigational Site Number 752001, Stockholm